CLINICAL TRIAL: NCT02472652
Title: An Open-label Study to Determine the Effect of Switching to Aripiprazole Once Monthly for Subjects With Schizophrenia Experiencing Worsening Sexual Dysfunction With Invega Sustenna or Risperdal Consta
Brief Title: Aripiprazole, Abilify Maintena Collaborative Clinical Protocol
Acronym: KISS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of adequate enrollment
Sponsor: Gazda, Thomas D., M.D., PC (Individual)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COL.AOM.2013-007
Record Dates: First submitted 2015-06-10; First posted 2015-06-16 (Estimated); Results first posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-03

CONDITIONS: Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abilify Maintena (Other): Subjects will be switched to Abilify Maintena (Aripiprazole) LAI monthly doses of 400mg, 300mg, 200mg or 160mg and have their sexual functioning reevaluated over a 3 month period to determine if there is any significant sexual functioning improvement.
  Interventions: Drug: Abilify Maintena

INTERVENTIONS:
Drug: Abilify Maintena — For subjects who meet inclusion/exclusion criteria for this study a switch from Palliperidone Palmitate or Risperidone injectable will be made to Abilify Maintena for a 3 month period to determine if there are changes in sexual dysfunction ratings over this time period
  Other Names: Aripiprazole

SUMMARY:
Sexual dysfunction is highly prevalent in schizophrenic patients, affecting up to 80% of men and women. Antipsychotic induced sexual side effects may be a barrier to treatment compliance. Antipsychotics such as Risperdal Consta and Invega Sustenna are known to have higher rates of causing prolactin elevations that may be implicated in sexual dysfunction. The basic premise of this study is to identify patients who believe they have experienced sexual dysfunction on Risperdal Consta or Invega Sustenna and switch to the alternative long acting injectable antipsychotic, Abilify Maintena which tends to lower prolactin levels. Measures of sexual sexual functioning using the self rated 5 item Arizona Sexual Experience Scale (ASEX) as the primary outcome measure will be made over a 3 month period to determine if such a switch is helpful.

DETAILED DESCRIPTION:
The study will be performed at several sites and oversight of the study is being monitored by Thomas D Gazda MD PC in accordance with established research principals, the ICH GCP (International Conference on Harmonization Good Clinical Practice) Guideline, FDA regulations and applicable regulatory requirements and local laws.

Source documents will be used to help ensure that patients meet diagnostic criteria for schizophrenia.

All AE (Adverse Event) verbatim descriptions will be performed (investigator terms from the CRF, Clinical Research File) will be classified into standardized medical terminology using the Medical Dictionary for Regulatory Activities (MedDRA).

Treatment emergent AEs (TEAEs) will be summarized. The incidence of TEAEs will be reported as the number (percentage) of subjects with TEAs by SOC (Standard of Care) and PT (Preferred Term). The number(percentage) of subjects with TEAEs will also be summarized by relationship to study drug (possibly related, probably related and not related).

Adverse events will be summarized using the Safety Analysis Sets. The number of AEs and number and incidence (%) of subjects with AEs will be summarized by cohort or dose and overall. For clinically significant events, tome of onset and recovery will be reported.

The number (percentage) of subjects with TEAEs leading to death will be summarized by MedDRA SOC and PT. A subject data listing of all AEs leading to death will be provided.

The number(percentage) of subjects with SAEs will be summarized by MedDRA SOC and PT.

The number (percentage) of subjects with TEAEs leading to discontinuation from study drug will be summarized by MedDRA SOC and PT. A subject data listing of all AEs leading to discontinuation from the study will be provided.

All safety analysis will be performed on the Safety Analysis Sets. Safety data will be summarized on an "as treated" basis using descriptive statistics (e.g. n, mean, standard deviation, median, minimum, maximum, for continuous variables: n(%) for categorical variables). Safety variables include TEAEs, clinical laboratory parameters, vital signs, SST). Study Day 1 for all safety analysis will be defined as the date of the first dose of study drug.

The primary analysis of the primary efficacy endpoint will be based on a one-sample two sided t-test. Missing values will be imputed using the last observation carried forward (LOCF). The ASEX at the end of the 3 months of treatment is considered to be lower than baseline if the 2-sided p-value of the one-sample t-test statistic is less than or equal to 0.05. As additional information, the two-sided 95% confidence interval for the change from baseline in ASEX score will be provided based on t-distribution at the end of the 3 months of aripiprazole once monthly treatment and at each scheduled visit.

As sensitivity analysis, the primary analysis will be repeated based on the observed data; also, a mixed effect analysis of covariance regression will be used to model the change from baseline in ASEX at scheduled visits. Baseline ASEX scores will be the fixed effect, subject will be the random effect, and scheduled visit will be the repeated factor in the model.

The key secondary analysis will be analyzed in the same way as the primary efficacy analysis

The study -conduct duration is approximately 4 months. Screening for subjects will last approximately 8 months for a total study duration of 12 months.

it is projected that a minimum of 22 subjects will be enrolled with an estimate that 19 subjects will complete the study.

ELIGIBILITY:
Inclusion Criteria:

1. Are able to provide written informed consent
2. Have a primary diagnosis of schizophrenia as determined by DSM-IV or DSM-V criteria.
3. Have a history of schizophrenia for greater than or equal to 2 years prior to screening documented from a reliable source (e.g. healthcare provider or medical records), and a history of symptom exacerbation or relapse when not receiving antipsychotic treatment
4. Are currently taking Invega Sustenna or Risperdal Consta
5. Have sexual dysfunction as defined by a score of greater than or equal to 19 on the ASEX or a score of greater than or equal to 5 on any one of item or a score of greater than or equal to 4 on any of each of three items (total score greater than or equal to 12 on the three items)
6. Experienced sexual dysfunction while treated with Invega Sustenna or Risperdal Consta
7. Have a minimal baseline sexual activity as defined as an ASEX score recalled from prior to initiation of Invega Sustenna or Risperdal Consta that is at least 2 points less than the total score at screening and not greater than or equal to 25 in severity.
8. Are able to understand the nature of the study and follow protocol requirements, including the prescribed dosage regimens, IM depot injection, discontinuation of prohibited concomitant medications, read and understand the written word in order to complete subject-reported outcome measures (including sexual functioning), and be reliably rated on assessment scales
9. Are male or female subjects who are surgically sterile or willing to employ a form of birth control including vaginal diaphragm, intrauterine device, birth control pill, birth control implant, birth control once monthly injections, condom or vaginal sponge with spermicide.

Exclusion Criteria:

1. Are female with amenorrhea for 3 consecutive months prior to screening, with the exception of women who are on Depo-Provera or oral contraceptives for the purpose of suppressing menstruation
2. Has a current DSM-IV or DSM-V diagnosis other that schizophrenia including schizophreniform disorder, schizoaffective disorder, major depressive disorder, bipolar disorder, delirium, dementia, amnestic or other cognitive disorders. Also excluded are subjects with borderline, paranoid, histrionic, schizotypal, schizoid, antisocial personality disorder, or any Axis II disorders or confounding Axis I disorders.
3. Has a CGI-S score at screening of grater than or equal to 5 (i.e. markedly ill or greater)
4. Has a diagnosis of type I or Type II diabetes unless diet controlled
5. Uses more than once daily antihypertensive medication, or greater than once per day dosing is allowed if on monotherapy (e.g. angiotensin-converting-enzyme inhibitors, angiotensin II receptor blockers, alpha blockers, and calcium channel blockers) with the exception of beta blockers and diuretics which are only allowed if once per day.
6. Is considered resistant or refractory to antipsychotic treatment by history (failed two prior antipsychotic medication studies) or response only to clozapine -

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12-31 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Gazda, MD, Principal Investigator — Private Practice
Locations (1):
- Mohammed Ramadan MD Private Practice, Bullhead City, Arizona, United States

REFERENCES:
- [Background] Baggaley M. Sexual dysfunction in schizophrenia: focus on recent evidence. Hum Psychopharmacol. 2008 Apr;23(3):201-9. doi: 10.1002/hup.924. PMID 18338766
- [Background] Henderson DC, Doraiswamy PM. Prolactin-related and metabolic adverse effects of atypical antipsychotic agents. J Clin Psychiatry. 2008;69 Suppl 1:32-44. PMID 18484806
- [Background] Hanssens L, L'Italien G, Loze JY, Marcus RN, Pans M, Kerselaers W. The effect of antipsychotic medication on sexual function and serum prolactin levels in community-treated schizophrenic patients: results from the Schizophrenia Trial of Aripiprazole (STAR) study (NCT00237913). BMC Psychiatry. 2008 Dec 22;8:95. doi: 10.1186/1471-244X-8-95. PMID 19102734
- [Result] de Boer MK, Wiersma D, Bous J, Sytema S, van der Moolen AE, Wilffert B, Hamamura T, Knegtering H. A randomized open-label comparison of the impact of aripiprazole versus risperidone on sexual functioning (RAS study). J Clin Psychopharmacol. 2011 Aug;31(4):523-5. doi: 10.1097/JCP.0b013e318222bb29. No abstract available. PMID 21720224

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abilify Maintena
Started | 2
Completed | 1
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Abilify Maintena
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2
ASEX (Arizona Sexual Experiences Scale) [Number; unit: units on a scale] — ASEX (Arizona Sexual Experiences Scale) score at baseline and end of study. This is a five item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm and satisfaction from orgasm. possible total scores range from 5 to 30, with the higher scores indicating more sexual dysfunction. Population: Second subject lost to follow up
  units on a scale
    number analyzed (Participants) | 1
    (all) | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Arizona Sexual Experiences Scale (ASEX) Score
Description: Subjects enrolled in this study will be followed for an average of about 5 months. The ASEX will be done at screening to ensure subjects meet criteria for sexual dysfunction as defined by the scale. In addition subjects must remember at least a 2 point change in the scale since starting Invega Sustenna or Risperdal Consta. Subjects must also score no greater than or equal to 25 on the scale to ensure a baseline of minimal sexual activity. The primary outcome of the study is the change in ASEX score from Baseline to Endpoint. Total scores range from 5 - 30 with the higher scores indicating more sexual dysfunction.
Time Frame: Baseline and 12 weeks
Population: Data no available for Subject 2 as lost to follow up
Measure: Number; unit: units on a scale
Arm/Group | Abilify Maintena
Number analyzed (Participants) | 1
units on a scale | 11

2. Secondary Outcome: Prolactin Concentrations ng/ml (Normal Range 4.0 - 15.2ng/ml)
Description: Subjects enrolled in this study will be followed for an average of about 5 months. Serum prolactin concentrations will be measured to assess change from Baseline to Endpoint
Time Frame: Baseline and Endpoint average of about 5 months
Population: Subject 2 not analyzed as lost to follow up
Measure: Number; unit: ng/ml
Arm/Group | Abilify Maintena
Number analyzed (Participants) | 1
ng/ml
  Baseline | 49.2
  5 months | 14.2
Statistical Analysis 1: Comparison: Abilify Maintena; Test type: Other; change in prolactin = 30

ADVERSE EVENTS:
Arm/Group | Abilify Maintena
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abilify Maintena (N=2)
hospitalization (Psychiatric disorders) | 1 (1) — subject hospitalized and lost to follow up after an apparent overdose
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abilify Maintena (N=2)
urinary retention (Renal and urinary disorders) | 1 (1) — only adverse event reported was 2nd subject reported difficulty urinating at visit 5 then lost to follow up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes